CLINICAL TRIAL: NCT05015907
Title: Ultrasound-guided Selective Supraclavicular Nerve Block for Postoperative Pain Control in Pediatric Patients Receiving Hickman Catheter, Chemoport or Perm Cath Insertion : a Randomized Controlled Trial
Brief Title: Ultrasound-guided Selective Supraclavicular Nerve Block for Postoperative Pain Control in Pediatric Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-2105-150-1222
Record Dates: First submitted 2021-08-05; First posted 2021-08-23 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Cancer Pediatric
Keywords: selective supraclavicular nerve block; postoperative pain control; Hickman catheter; chemoport; Perm cath
MeSH Terms: conditions — Neoplasms | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Selective supraclavicular nerve block (Experimental): After induction of anesthesia, the anesthesiologist sterilizes the skin of the area to be punctured. In the test group, an Ultrasound-guided selective supraclavicular nerve block is performed using 0.5% Ropivacaine 0.1mL/kg (Maximum dose: 5mL).
  Interventions: Drug: Ropivacaine
- Control (Active Comparator): The nerve block is not performed in the control group.
  Interventions: Other: Control (without intervention)

INTERVENTIONS:
Drug: Ropivacaine — The nerve involved in the operation of Hickman catheter, chemoport, and Perm cath is the supraclavicular nerve. Therefore, it is judged that if only this nerve is selectively blocked, pain control can be effectively performed with a small amount of local anesthetic, and relatively few side effects occur.
  Arms: Selective supraclavicular nerve block
Other: Control (without intervention) — No intervention
  Arms: Control

SUMMARY:
This prospective randomized controlled trial aims to investigate the effect of ultrasound-guided selective supraclavicular nerve block on pain control after Hickman catheter, chemoport, or Perm cath insertion in children.

DETAILED DESCRIPTION:
Pediatric patients undergoing surgical insertion of a Hickman catheter, chemoport, or Permcath are randomly assigned to a test group (Ultrasound-guided selective supraclavicular nerve block with Ropivacaine) and a control group (Nerve block is not performed).

Immediately after induction of general anesthesia, in the test group, the supraclavicular nerve block was selectively performed using ultrasound using 0.1mL/kg of 0.5% Ropivacaine (Maximum dose: 5mL), and the nerve block was not completed in the control group. After that, a Hickman catheter, chemoport, or Permcath is surgically inserted in the usual way and allowed to recover from anesthesia.

The pain score is evaluated between 10 and 30 minutes of entering the recovery room (1 hour after the procedure) and 1 hour, 3 hours, and 24 hours after leaving the recovery room by another research team who is unaware of the group assignment. In addition, the use of additional analgesic drugs and related side effects were collected before discharge.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients receiving Hickman catheter, chemoport, or Perm cath implantation (3 years ≤, <18 years)
* One or more of the parents (or guardians), after hearing and understanding a sufficient explanation about this clinical trial, decides to participate voluntarily and agrees in writing to abide by the precautions
* In the case of a study subject aged seven years or older, a person who voluntarily decides to participate in this clinical trial and agrees in writing to abide by the precautions after hearing and understanding a sufficient explanation about this clinical trial

Exclusion Criteria:

* Patients who undergo surgery other than the surgery.
* Patients with diseases whose sensitivity to pain is different from that of the general public
* Unstable vital signs (heart rate, blood pressure)
* General contraindications of Ropivacaine
* Patients with a history of allergy to opioids
* Severe renal dysfunction (Creatinine> 3.0 mg/dl)
* Severe liver dysfunction (aspartate transaminase > 120 unit/L, alanine aminotransferase > 120 unit/L)
* Peripheral nervous system abnormalities
* At risk of malignant hyperthermia
* Other cases that the researcher judges to be inappropriate

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2021-10-22 (Actual); Primary Completion 2023-02-23 (Actual); Study Completion 2023-02-24 (Actual)

PRIMARY OUTCOMES:
Pain score | Pain score measured when communication is possible between 10 and 30 minutes after entering the recovery room.
  Wong-Baker Faces Pain Rating Scale is used
Pain score | Pain score measured when communication is possible between 10 and 30 minutes after entering the recovery room.
  Numeric rating scale is also evaluated if communication is possible

SECONDARY OUTCOMES:
Pain score | Pain score for 1 hour, 3 hours, and 24 hours after leaving the recovery room
  Wong-Baker Faces Pain Rating Scale is used
Pain score | Pain score for 1 hour, 3 hours, and 24 hours after leaving the recovery room
  Numeric rating scale is also evaluated if communication is possible
Additional narcotic analgesics administered | Within 24 hours of the end of surgery
  Amount per body weight of additional narcotic analgesics administered.
Additionally administered non-narcotic analgesics | Within 24 hours of the end of surgery
  Amount per body weight of additionally administered non-narcotic analgesics.
Side effects related to pain medication | Within 24 hours of the end of surgery
  Nausea, Vomit, Constipation, Pruritus, Dizziness, Dry mouth, Sedation, etc.
Complications related to ropivacaine use | Within 1 hour after procedure
  Arrhythmia, Hypotension, ST change, Dizziness, Convulsion, etc.
Whether diaphragmatic palsy | Within 24 hours of the end of surgery
  It is confirmed by chest X-ray taken in the operating room. Diaphragmatic palsy can usually be suspected on chest X-rays showing abnormal hemidiaphragm elevation. Therefore, we will check the chest X-ray for abnormal hemidiaphragm elevation.
Whether diaphragmatic palsy | Within 24 hours of the end of surgery
  It is confirmed by lung ultrasound in the recovery room. Hemidiaphragm visualization by ultrasound is achieved from an anterior approach, with the patient in a supine position.
  At the ultrasound, the diaphragm appears as a thick echogenic line. M-mode US may be used to measure the direction of diaphragmatic motion and the amplitude of excursion.
  The two indexes usually used for the diagnosis of diaphragmatic paralysis include a Tdi value <2 mm and a diaphragm thickening fraction (TFdi)value <20% [Tdi: The thickening of the diaphragm, TFdi: (thickness at the end of the inspiration - thickness at the end of expiration)/thickness at the end of expiration (in %)].
Hospital stay | No more than one month
  The period from discharge from recovery room to discharge
Check the blockage | When communication is possible between 10 and 30 minutes after entering the recovery room.
  The quality of the selective supraclavicular nerve block will be tested with loss of cold sensation using an alcohol swab.

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Tae Kim, MD,PhD, Principal Investigator — Seoul National University Hospital, Seoul National University College of Medicine
Locations (1):
- Jin-Tae Kim, Seoul, South Korea

REFERENCES:
- [Derived] Park JB, Song IS, Kang PY, Ji SH, Jang YE, Kim EH, Lee JH, Kim HS, Kim JT. Ultrasound-guided selective supraclavicular nerve block for postoperative pain control in children receiving Hickman catheter or chemoport insertion: A randomized controlled trial. Paediatr Anaesth. 2024 Jan;34(1):35-41. doi: 10.1111/pan.14745. Epub 2023 Aug 16. PMID 37587734